CLINICAL TRIAL: NCT01546129
Title: Effect of Dianatal Obstetric Gel (Cross-linked Polyacrylic Acid) on Outcomes in Vaginal Delivery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, boris kaplan, Prof. Boris Kaplan, Rabin Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: DOCS001
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-01

CONDITIONS: Labor, First Stage; Labor, Second Stage

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Dianatal Obstetric Gel (Experimental): Standard of care according to the established Guidelines of the Department plus use of Dianatal applied with a vaginal applicator in stage I and stage II of labor
  Interventions: Device: Dianatal Obstetric Gel (Cross-linked polyacrylic acid)
- Control (No Intervention): Standard of care according to the established Guidelines of the Department.
  Interventions: Device: Dianatal Obstetric Gel (Cross-linked polyacrylic acid)

INTERVENTIONS:
Device: Dianatal Obstetric Gel (Cross-linked polyacrylic acid) — Dianatal (approx. 30 mL in total) will be intermittently administered to the birth canal after vaginal examination in labor using the Dianatal applicator or the syringe or the fingers. Dianatal Stage I is used during labor stage I, Dianatal Stage 2 is used during stage 2. After rupture of the membranes supplementary Dianatal is applied within 5 to 20 minutes.

SUMMARY:
Perineal massage at the end of labor stage 2 has been investigated in 2 randomized controlled trials using a water soluble lubricant. In one trial a significant reduction of labor stage 2 has been found, both trials did not show a significant increase of perineum integrity.

In the HCB Swiss Study both a significant reduction of labor stage 2 by 30 % as well as a significant increase of perineal integrity have been shown. No adverse events have been reported.

(see also Obstetric gel shortens second stage of labor and prevents perineal trauma in nulliparous women: a randomized controlled trial on labor facilitation. Schaub AF, Litschgi M, Hoesli I, Holzgreve W, Bleul U, Geissbuhler V. J Perinat Med 2008; 36 (2): 129-135).

Today's practice- Lubricants are widely used to enable manual vaginal examination during labor. In Israel midwifes are using Almond Oil for perineal massage at the end of labor stage 2 to protect the perineum. It has been shown for the first time that the use of the Dianatal Obstetric Gel facilitates vaginal childbirth in humans. Dianatal has been introduced to the EU markets in 2008.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age between 18 and 40 years
* signed written informed consent,
* intention for vaginal delivery,
* nulliparous state or multiparous state
* singleton baby in vertex presentation
* estimated birth weight between 1500 g and 4500 g
* low risk pregnancies at term and late preterm (34 to 42weeks of gestational age)

Exclusion Criteria:

* contraindications for vaginal delivery
* indications for an amnion infection syndrome
* suspect for fetal malformations
* indications for cephalopelvic disproportion
* severe concomitant diseases of the mother

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-04; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Effects on c-section rates
Effects on vaginal operative intervention rates (forceps, vaccum)
Effects on prolonged second stage
Effects on vaginal and Perineum: tears
Effect on episiotomy rate
Effect on labor outcome in premature infants

SECONDARY OUTCOMES:
Effect on labor duration stage 2 (full dilatation of the cervix until delivery of the baby).
Effect on labor duration stage 1 (cervical dilatation of uterus between 4 cm and 10 cm, the beginning of stage 1, i.e. 4 cm dilatation should be evaluated as close as possible within routine examination periods)
Effect on birth trauma (birth canal lacerations): vaginal lesions, perineal lesions
Effect on labor outcomes in state after c-section
Effect on pain experience (pain reduction) measured by visual analog scale: use of epidural
Effect on postpartum vaginal or urethral burn feeling
Effect on newborn outcomes (APGAR score 1, 5 and 10 min after birth; umbilical cord pH; reduction of newborn trauma)

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel